CLINICAL TRIAL: NCT06983743
Title: A Phase 1 First-in-Human Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of ERAS-0015 Monotherapy and in Combination in Patients Advanced Solid Tumors
Brief Title: A Study of ERAS-0015 in Patients With Advanced or Metastatic Solid Tumors
Acronym: AURORAS-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-0015-01
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Solid Tumors
Keywords: Solid Tumor; Advanced Solid Tumor; solid malignancies; Targeted therapy; Molecular alterations; pembrolizumab; Keytruda; panitumumab; Vectibix; Metastatic Solid Tumor; Neoplasms
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — pembrolizumab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ERAS-0015 Monotherapy Dose Optimization. (Experimental): Escalating doses of ERAS-0015 administered orally.
  Interventions: Drug: ERAS-0015
- ERAS-0015 Combination Dose Optimization (Experimental): ERAS-0015 administered orally with another investigational agent.
  Interventions: Drug: ERAS-0015 in combination

INTERVENTIONS:
Drug: ERAS-0015 — ERAS-0015 Administered orally
  Arms: ERAS-0015 Monotherapy Dose Optimization.
Drug: ERAS-0015 in combination — ERAS-0015 Administered orally and in combination with either Keytruda (pembrolizumab) via IV administration or Vectibix (panitumumab) via IV administration.
  Other Names: Pembrolizumab; Keytruda; Panitumumab; Vectibix
  Arms: ERAS-0015 Combination Dose Optimization

SUMMARY:
The main purpose of the study is to assess whether the study drug, ERAS-0015, is safe and tolerable when administered to patients with advanced or metastatic solid tumors with certain RAS mutations. ERAS-0015 will be given alone or in combination with other treatments.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1/1b, open-label, multicenter clinical study of ERAS-0015 as a monotherapy and in combination with other cancer therapies. The study will commence with dose optimization of ERAS-0015 monotherapy, followed by dose optimization of ERAS-0015 in combination with other cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing and able to give written informed consent
* Pathological documentation of tumor type and mutation prior to the first dose of study drug(s), for applicable cohorts.
* There is no available standard systemic therapy available for the patient's tumor histology and/or molecular biomarker profile; or standard therapy is intolerable, not effective, or not accessible; or patient has refused standard therapy
* Able to swallow oral medication
* Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Adequate cardiovascular, hematological, liver, and renal function
* Willing to comply with all protocol-required visits, assessments, and procedures

Exclusion Criteria:

* Previous treatment with a RAS inhibitor
* Is currently receiving another study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of the first dose of ERAS-0015
* Received prior palliative radiation within 14 days of Cycle 1, Day 1
* Have primary central nervous system (CNS) tumors
* Prior surgery (e.g., gastric bypass surgery, gastrectomy) or gastrointestinal dysfunction (e.g., Crohn's disease, ulcerative colitis, short gut syndrome) that may affect drug absorption
* Have any underlying medical condition, psychiatric condition, or social situation that, in the opinion of the Investigator, would compromise study administration as per protocol or compromise the assessment of AEs
* Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Study Day 1 up to Day 21
  Based on toxicities observed
Maximum tolerated dose (MTD) | Study Day 1 up to Day 21
  Based on toxicities observed
Recommended dose for expansion (RDE) | Study Day 1 up to Day 21
  Based on toxicities observed
Adverse Events | Study Day 1 up to Day 21
  Incidence and severity of treatment-emergent AEs and serious AEs
Plasma concentration (Cmax) | Study Day 1 up to 65
  Maximum plasma concentration of ERAS-0015
Time to achieve Cmax (Tmax) | Study Day 1 up to 65
  Time to achieve maximum plasma concentration of ERAS-0015
Area under the curve | Study Day 1 up to 65
  Area under the plasma concentration-time curve of ERAS-0015
Half-life | Study Day 1 up to 65
  Half-life of ERAS-0015

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Time to Response (TTR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Gerri Lee, Study Director — Erasca, Inc.
Locations (5):
- United States (5):
  - Florida Cancer Specalists, Sarasota, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas at Tyler, Tyler, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No